CLINICAL TRIAL: NCT02451995
Title: A Prospective Multi-centre Study of Effectiveness of Ripple Mapping for Atrial Tachycardia Ablation
Brief Title: Effectiveness of Ripple Mapping in Atrial Tachycardia Ablation
Acronym: RIPPLE-AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14HH2319
Record Dates: First submitted 2015-04-14; First posted 2015-05-22 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Atrial Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ripple Mapping guided AT ablation (Experimental): Ripple Mapping (Imperial College) software (Biosense Webster) will be used to diagnose the mechanism of AT and guide ablation
  Interventions: Device: Ripple Mapping guided AT ablation
- Local activation Time Mapping AT Ablation (Active Comparator): Standard activation mapping will be used to guide ablation.
  Interventions: Device: Local activation Time Mapping AT Ablation

INTERVENTIONS:
Device: Ripple Mapping guided AT ablation — Diagnosing the mechanism and delivering ablation within the atria in patients with atrial tachycardia on the basis of Ripple Mapping
  Arms: Ripple Mapping guided AT ablation
Device: Local activation Time Mapping AT Ablation — Diagnosing the mechanism and delivering ablation within the atria in patients with atrial tachycardia on the basis of local activation time mapping
  Arms: Local activation Time Mapping AT Ablation

SUMMARY:
Tachycardia's (fast heart rhythms) can lead to troublesome palpitations, dizziness, blackouts and breathlessness. They are caused either by a cluster of abnormal cells within the heart, or an electrical short circuit which rotates rapidly around the heart. Sometimes these can be controlled with tablets, though owing to side effects many patients want something else. Many tachycardia's can be cured by a procedure known as an "ablation". In essence, either the focus of abnormal cells or the narrowest point of the short circuit causing the abnormal heart rhythm (the source) is electrically destroyed (burnt) resulting in restoration of the normal heart beat.

One form of tachycardia is known is Atrial Tachycardia (AT). These arise from the top two chambers of the heart (the atrium). Interestingly, this problem is frequently seen in patients who have previously undergone an ablation or surgical procedure for a condition called Atrial Fibrillation. In others the reason for its occurrence is unknown. Current strategies to find the "source" during an ablation procedure are technically challenging resulting in long procedure times. Sometimes the wrong source is found resulting in ablation at the incorrect site.

Ripple Mapping (RM) is a novel system that Investigators at Imperial College are looking to study. RM displays electrical information within the heart as a series of bars coming out of the chamber, with each bar representing signals travelling down the heart. By seeing the pattern of electrical information, they believe it will show the pattern of the tachycardia better than conventional techniques. In a previous retrospective study that they conducted, RM found the source of the tachycardia in 80% of the maps, compared to only 50% with the current system. Investigators at Imperial College have identified why they did not get 100% and they believe that, in future, RM will find the source of the tachycardia first time, and every time.

DETAILED DESCRIPTION:
Conventional mapping strategies used to find the "source" of "atrial tachycardia" within the heart are technically challenging resulting in long procedure times. Sometimes the wrong source is found resulting in ablation at the incorrect site.

In a retrospective study conducted by investigators at Imperial College, Ripple Mapping (RM) found the source of the tachycardia 80% of the time, compared to only 50% with conventional maps (known as local activation time maps). They have since studied the reasons why did not achieve 100%, but could not improve matters with a retrospective data-set. They believe that, in future, Ripple mapping will find the source of the tachycardia first time, and every time. The purpose of this study is to prospectively test whether Ripple Mapping is better at finding the source of the "atrial tachycardia" (AT) than conventional local activation time mapping.

Patients referred for clinically indicated AT ablation by their electro-physiologist will be recruited. For each patient recruited to the study, they will be block randomized into 2 arms: Ripple Mapping guided AT ablation, or Conventional AT guided Ablation (local activation time mapping). Following explanation of the study the patients will be allowed time to decide on whether they would like to participate.

Following completion of the consent procedure the patient will undergo the electrophysiology study as is routine standard practice. This is usually performed by inserting plastic tubes (catheters) into the heart using the vessels in the groin. Once the catheter is in the atrium (top chambers of the heart) the catheter will be moved to different locations in the chamber to gather the electrical information of the tissue. Using "CARTO3v4 ConfiDENSE", a 3-Dimensional map of the geometry of the heart chambers will be constructed.

Patient randomized to RM will proceed as follows: Once sufficient points have been collected, the Ripple Map will be played in order to diagnose the source of the tachycardia. In the context of a clear diagnosis, the operator can proceed to ablation at the defined source from the Ripple map. Termination of the tachycardia with ablation will be used to confirm the diagnosis was correct. A single entrainment is permissible where the diagnosis is unclear.

Patients randomized to conventional local activation time (LAT) mapping will proceed according to standard practice of the operator. When the operator is satisfied adequate number of points have been collected, the operator can proceed to ablation if the diagnosis is clear. A single entrainment is permissible where the diagnosis is unclear. The endpoints measured will include:

1. Tachycardia change or termination following first series of ablations with Ripple Mapping vs local activation time mapping.
2. The reliance on entrainment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing clinically indicated ablation for atrial tachycardia using 3D mapping.

Exclusion Criteria:

1. Patients with typical flutter.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, MBBChir PhD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linton NW, Koa-Wing M, Francis DP, Kojodjojo P, Lim PB, Salukhe TV, Whinnett Z, Davies DW, Peters NS, O'Neill MD, Kanagaratnam P. Cardiac ripple mapping: a novel three-dimensional visualization method for use with electroanatomic mapping of cardiac arrhythmias. Heart Rhythm. 2009 Dec;6(12):1754-62. doi: 10.1016/j.hrthm.2009.08.038. Epub 2009 Sep 3. PMID 19959125
- [Background] Jamil-Copley S, Linton N, Koa-Wing M, Kojodjojo P, Lim PB, Malcolme-Lawes L, Whinnett Z, Wright I, Davies W, Peters N, Francis DP, Kanagaratnam P. Application of ripple mapping with an electroanatomic mapping system for diagnosis of atrial tachycardias. J Cardiovasc Electrophysiol. 2013 Dec;24(12):1361-9. doi: 10.1111/jce.12259. Epub 2013 Oct 10. PMID 24118203
- [Derived] Luther V, Agarwal S, Chow A, Koa-Wing M, Cortez-Dias N, Carpinteiro L, de Sousa J, Balasubramaniam R, Farwell D, Jamil-Copley S, Srinivasan N, Abbas H, Mason J, Jones N, Katritsis G, Lim PB, Peters NS, Qureshi N, Whinnett Z, Linton NWF, Kanagaratnam P. Ripple-AT Study: A Multicenter and Randomized Study Comparing 3D Mapping Techniques During Atrial Tachycardia Ablations. Circ Arrhythm Electrophysiol. 2019 Aug;12(8):e007394. doi: 10.1161/CIRCEP.118.007394. Epub 2019 Aug 9. PMID 31394921

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 were excluded. This was due premature termination of AT whilst mapping (n=6), AT non-inducibility (n=9), or degeneration to alternating ATs/atrial fibrillation prior to the delivery of ablation (n=4). Left atrial appendage thrombus on Trans Oesophageal Echo seen at the start of the procedure (n=3) resulted in immediate procedural cessation.
Groups:
- Conventional Local Activation Time Mapping Ablation: Standard activation mapping will be used to guide ablation.
  Conventional AT ablation: Diagnosing the mechanism and delivering ablation within the atria in patients with atrial tachycardia on the basis of activation mapping
Period: Overall Study
Arm/Group | Ripple Mapping Guided AT Ablation | Conventional Local Activation Time Mapping Ablation
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conventional AT Ablation: Standard activation mapping and entrainment will be used to guide ablation.
  Conventional AT ablation: Diagnosing the mechanism and delivering ablation within the atria in patients with atrial tachycardia on the basis of activation mapping and entrainment
- Total: Total of all reporting groups
Arm/Group | Ripple Mapping Guided AT Ablation | Conventional AT Ablation | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 65 (10) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data not collected Population: Gender data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: A Composite of the Total Number of Participants With Either Tachycardia Change or Tachycardia Termination With First Ablation Set.
Description: The total number of participants in each arm with either a change of termination of their atrial tachycardia following delivery of the first ablation set post map categorisation.
Time Frame: Participants will be followed for the duration of hospital stay (typically an overnight stay, hence 24hrs.
Measure: Count of Participants; unit: Participants
Groups:
- Conventional AT Ablation: Standard activation mapping will be used to guide ablation.
  Conventional AT ablation: Diagnosing the mechanism and delivering ablation within the atria in patients with atrial tachycardia on the basis of activation mapping
Arm/Group | Ripple Mapping Guided AT Ablation | Conventional AT Ablation
Number analyzed (Participants) | 42 | 41
Participants | 38 | 29

ADVERSE EVENTS:
Time Frame: 24hrs
Arm/Group | Ripple Mapping Guided AT Ablation | Conventional AT Ablation
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT02451995/Prot_SAP_000.pdf